CLINICAL TRIAL: NCT01173016
Title: Pilot Study of Administration of Intravenous Laronidase Following Allogeneic Transplantation for Hurler Syndrome
Brief Title: Administration of IV Laronidase Post Bone Marrow Transplant in Hurler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS090; MT2009-20 (Other: Blood and Marrow Transplantation Program); 1004M80513 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Hurler Syndrome
Keywords: mucopolysaccharide IH (MPS IH)
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laronidase After Transplantation (Experimental): Patients with Mucopolysaccharidosis type IH (MPS I, Hurler syndrome) treated with a prior allogeneic transplant >2 years previously and treated with Laronidase weekly for 2 years after transplant.
  Interventions: Drug: Laronidase

INTERVENTIONS:
Drug: Laronidase — Laronidase 0.58 mg/kg intravenously (IV) once a week for a maximum of 2 years
  Other Names: Aldurazyme

SUMMARY:
This is a single center pilot study in which Laronidase will be given weekly for two years in patients with Hurler syndrome, also known as mucopolysaccharide IH (MPS I, Hurler syndrome), that have previously been treated with an allogeneic transplant.

DETAILED DESCRIPTION:
This 2-year open-label pilot study of laronidase includes patients (age 5-13 years) who are at least 2 years post-hematopoietic cell transplantation (HCT) and donor engrafted. Outcomes are assessed semi-annually and compared to historic controls. Eligible patients will receive Laronidase as an infusion over several hours once a week at a local site. The dosing of enzyme will be the standard doses recommended by Genzyme.

The findings of this Pilot Study will be used to assess whether a subsequent larger study can be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Mucopolysaccharidosis type IH (MPS I, Hurler syndrome) treated with a prior allogeneic transplant >2 years previously
* Age <14 years old
* >10% engrafted based on recent testing (<4 months prior to enrollment)
* Willing to commit to traveling to the University of Minnesota every 6 months
* Written informed consent prior to the performance of any study related procedures

Exclusion Criteria:

* Previous administration of Laronidase enzyme > 3 months post transplantation
* Anticipated survival less than 2 years
* History of cardiac or pulmonary insufficiency, including an ejection fraction (EF) < 40% or those requiring continuous supplemental oxygen

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2016-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Lund TC, Miller WP, Liao AY, Tolar J, Shanley R, Pasquali M, Sando N, Bigger BW, Polgreen LE, Orchard PJ. Post-transplant laronidase augmentation for children with Hurler syndrome: biochemical outcomes. Sci Rep. 2019 Oct 1;9(1):14105. doi: 10.1038/s41598-019-50595-1. PMID 31575939
- See also: Related Info — https://www.nature.com/articles/s41390-019-0541-2
- See also: Related Info — https://www.nature.com/articles/s41598-019-50595-1#citeas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laronidase After Transplantation
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adherence to the Scheduled Weekly Infusion by the Participants
Description: To determine the feasibility of giving weekly Laronidase for 2 years in patients with Hurler syndrome after allogeneic transplantation, compliance throughout the study with drug administration, the percentage of adherence to the scheduled weekly infusion for each participant is measured.
Time Frame: 24 months
Measure: Median (Full Range); unit: percentage
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 10
percentage | 99 [79 to 100]

2. Primary Outcome: Number of Participants Experiencing Severe Adverse Events
Description: Number of participants experiencing severe adverse events that occur after administration with Laronidase to determine the feasibility of giving weekly Laronidase
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 11
Participants | 1

3. Secondary Outcome: Changes in Growth Velocity
Description: difference between baseline and month 24 growth velocities
Time Frame: Baseline, Month 24
Population: Baseline growth velocity value was available in six of ten participants. One female participant was excluded from the within-group growth analyses due to a bone age of 14.5 years
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 5
cm/year | -1.1 (3.8)

4. Secondary Outcome: Change in Muscle Strength
Description: Handgrip strength is measured three times in both hands with a mechanical handheld Biodex System 3 dynamometer (Biodex medical Systems, Inc., Shirley, NY) with the subject in a seated position at each visit; the average for each hand is presented.
Time Frame: Assessed from baseline every 6 months through 2 years; change between baseline and 24 months reported.If baseline and/or 24-month data were not available, the longest interval between measurements was reported, with a minimum requirement of 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 10
kg | 1.1 (1.9)

5. Secondary Outcome: Change in Peak Heart Rate to Monitor "Fitness"
Description: A modified Balke Treadmill Test was performed. Briefly, patients began walking at 2.0 mph with a 2% increase in grade every 2 min. A 12-lead electrocardiogram was monitored continuously throughout the test for the determination of heart rate and dysrhythmias or ischemic changes. Heart rate was measured at the end of each stage (i.e. every 2 min) .
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 10
bpm | 23 (18)

6. Secondary Outcome: Number of Participants Showing Improvements in Joint Range of Motion (ROM)
Description: Bilateral shoulder flexion, elbow extension, and hip extension were measured using goniometry. Improvements are defined for all joints as >5°.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 10
Participants
  Left or right shoulder ROM improvement | 4
  Left or right elbow ROM improvement | 3
  Left or right hip ROM improvement | 5

7. Secondary Outcome: Shortening Fraction to Determine Systolic Cardiac Function
Description: Cardiac ultrasounds were obtained at baseline and month 24. Two-dimensional imaging was obtained for determination of anatomy. Shortening fraction (SF [normal > 27%]) was calculated by standard methods to determine the normal systolic cardiac function
Time Frame: Baseline and month 24
Population: two subjects didn't have both baseline and month 24 echo data
Measure: Mean (Full Range); unit: percentage of systolic cardiac function
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 8
percentage of systolic cardiac function | 38 [34 to 52]

8. Secondary Outcome: Number of Participants With Changes in Cardiac Echo Structural Parameters
Description: Pulse-wave and color Doppler interrogation of cardiac valves was performed for determination of valve regurgitation
Time Frame: Baseline and month 24
Population: Two subjects didn't have both baseline and month 24 echo data
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 8
Participants
  Mitral regurgitation - unchaged | 7
  Mitral regurgitation - increased | 1
  Aortic regurgitation - unchanged | 5
  Aortic regurgitation - increased | 3

9. Secondary Outcome: Correlation of 6 Minute Walk Test With Anti-laronidase Antibody + Status
Description: 6 minute walk test (6MWT) was performed to assess overall physical function and health status. In brief, a 30m hospital corridor marked by colored tape at each end was used. Subjects were instructed to walk from end to end at their self-selected pace, while attempting to cover as much distance as possible in the 6 min. The patients were instructed to walk around the mark as they changed direction. The time and distance covered was recorded, as was the heart rate prior to and immediately after completion of the walk test.
  To find the association between the rate of change in 6MWT, and anti drug antibody (ADA) titer, a statistical test is performed adjusting for age at the time of enrollment.
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Laronidase After Transplantation
Number analyzed (Participants) | 10
meters | -14 [-28 to -1]
Statistical Analysis 1: Comparison: Laronidase After Transplantation; Impact of anti-laronidase antibody status on the change in 6MWT outcome was tested; Test type: Other; p = 0.038, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Laronidase After Transplantation
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laronidase After Transplantation (N=11)
Syncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laronidase After Transplantation (N=11)
Allergy Reaction/Hypersensitivity (Immune system disorders) | 1 (4)
Fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hives (Immune system disorders) | 1 (3)
Hypertension (Vascular disorders) | 3 (47)
Pain, Right Shoulder (General disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 3 (36)
Hypotension (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All listed serious and non-serious adverse events are infusion related except for a seizure that was thought to be unrelated to the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No